CLINICAL TRIAL: NCT01129934
Title: Pharmacological Anxiolysis With Promethazine as an Adjunctive Therapy for Acute Low Back Pain in the Adult Emergency Department
Brief Title: Morphine Versus Morphine-promethazine Combination for Acute Low Back Pain Relief in the Adult Emergency Department
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Halpern Pinchas, Chair, Department of Emergency Medicine, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-09-PH-701-CTIL
Record Dates: First submitted 2010-04-21; First posted 2010-05-25 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Low Back Pain
Keywords: Low Back Pain,; Emergency medicine,; Promethazine,; Morphine,; Pain relief
MeSH Terms: conditions — Low Back Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine-Promethazine (Experimental): Pain relief by administration of morphine-promethazine combination
  Interventions: Drug: Morphine-Promethazine
- morphine (Active Comparator): pain relief by administration of morphine
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: Morphine-Promethazine — administration of intravenous morphine 0.1mg/kg and promethazine 12.5 mg in a 500 Ml 0.9% saline
  Other Names: morphine-phenergan
  Arms: Morphine-Promethazine
Drug: morphine — Administration of intravenous morphine 0.1 mg/kg
  Other Names: morphine as a single drug
  Arms: morphine

SUMMARY:
Acute low back pain is a common cause for emergency department visits. Controversy remains regarding the optimal medication for acute low back pain relief. The investigators hypothesized that administration of pharmacological anxiolysis in addition to analgesia will improve pain relief and patient management in the emergency department.

DETAILED DESCRIPTION:
Acute low back pain is a common problem in the emergency department and pain relief is usually the first step in patients' management. Numerous medication options are available for acute LBP relief,each class of medication has its associated benefits and harms.Controversy remains regarding the optimal analgesic treatment.Anxiety has been found to be a predictive factor of pain intensity in patients with acute low back pain and anxiolysis by non-pharmacological measures has been shown to have a positive effect on pain management in the ED setting.

Promethazine is a first-generation H1 receptor antagonist of the phenothiazine chemical class used commonly as an antihistamine antiemetic. It has a strong anxiolytic-sedative effect and its safety and efficacy in managing anxiety related to medical procedures is well documented.It may be reasonable to assume that pharmacological anxiolysis with promethazine may assist in alleviation of acute pain in the strenuous environment of the ED.

ELIGIBILITY:
Inclusion Criteria:

1. An indication for opioid analgesia based in the ED (i.e. severe pain > 70mm on a 100mm VAS)
2. Age between 18-65 years
3. American Society of Anesthesiologists (ASA) score of 1 or 2, and no preexisting glaucoma, cardiac arrhythmia or pulmonary disease
4. Systolic blood pressure higher than 90 mmHg on admission
5. Willingness and ability to provide an informed consent
6. No known hypersensitivity to the medication used.

Exclusion Criteria:

1. Pregnant women
2. Patients who can not be under adult supervision following discharge from the emergency department.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Pain relief | Up to 24 hours (before analgesia administration and on discharge from the ED or admission to the hospital)
  Pain scores before and after treatment will be assessed on a 100mm VAS. The difference will be regarded as pain relief.

SECONDARY OUTCOMES:
Ambulatory status | Up to 24 hours (before analgesia administration and on discharge from the ED or admission to the hospital)
  Most patients who suffer from acute LBP are in severe pain and are unable to ambulate. The ambulatory status of every patient (e.g., able to walk independently, using a can, wheelchair, laying down and unable to sit or stand up)will be recorded before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pinchas Halpern, M.D, Study Chair — Tel-Aviv Medical Center, Tel-Aviv University, Israel
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel